CLINICAL TRIAL: NCT00282009
Title: Internet and Telephone Counseling for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000465179; R01CA104836 (NIH)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2014-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Basic Internet (Active Comparator): Basic Internet
  Interventions: Behavioral: Basic Internet
- Enhanced Internet (Experimental): Enhanced Internet
  Interventions: Behavioral: Enhanced Internet
- Enhanced Internet plus Phone (Experimental): Enhanced Internet + proactive telephone counseling
  Interventions: Behavioral: Enhanced Internet + phone

INTERVENTIONS:
Behavioral: Basic Internet — Basic Internet control intervention
  Arms: Basic Internet
Behavioral: Enhanced Internet — enhanced Internet cessation intervention
  Arms: Enhanced Internet
Behavioral: Enhanced Internet + phone — enhanced Internet plus proactive telephone counseling
  Arms: Enhanced Internet plus Phone

SUMMARY:
RATIONALE: Computer-assisted stop-smoking plans and telephone counseling may help people stop smoking. It is not yet known which computer-based smoking cessation program is more effective with or without telephone counseling in helping smokers quit smoking.

PURPOSE: This randomized clinical trial is studying two different computer-based smoking cessation programs to compare how well they work with or without telephone counseling in helping smokers quit smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of premium internet intervention vs premium internet with telephone intervention vs basic internet intervention, as determined by 7-day point prevalence abstinence at 12 months, in adult smokers.
* Compare the cost-effectiveness of these interventions in promoting smoking cessation.
* Determine the effects of internet-based interventions on measured use of the intervention (frequency and duration of use, utilization of behavioral coping, expert advices, and e-mail) in these patients.
* Determine the effects of internet-based interventions on variables important for behavior change including mediators (e.g., self-efficacy, use of internet social support) and moderators (e.g., gender, baseline motivation) of outcomes in these patients.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to gender and baseline motivation level. Patients are randomized to 1 of 3 intervention arms.

* Arm I (basic internet program): Patients are directed to a website of existing QuitNet™ smoking cessation materials. These materials are not tailored and have no interactive features.
* Arm II (premium internet program): Patients receive free 6-month access to the QuitNet™ website including interactive and individualized intervention features.
* Arm III (premium internet program plus telephone counseling): Patients receive free access to the QuitNet™ website as in arm II. Patients also receive up to 5 telephone counseling sessions, scheduled at their convenience.

All patients are assessed at baseline and then at 3, 6, 12, and 18 months.

PROJECTED ACCRUAL: A total of 2,205 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Smokes at least 5 cigarettes a day
* No prior use of QuitNet website
* Must have access to the internet and a telephone at home or work

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2205 (Actual)
Dates: Start 2004-08; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence as measured by 7-day point prevalence abstinence at 12 months following treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L. Graham, PhD, Principal Investigator — Lombardi Comprehensive Cancer Center
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graham AL, Bock BC, Cobb NK, Niaura R, Abrams DB. Characteristics of smokers reached and recruited to an internet smoking cessation trial: a case of denominators. Nicotine Tob Res. 2006 Dec;8 Suppl 1(Suppl 1):S43-8. doi: 10.1080/14622200601042521. PMID 17491170
- [Result] Graham AL, Papandonatos GD, Bock BC, Cobb NK, Baskin-Sommers A, Niaura R, Abrams DB. Internet- vs. telephone-administered questionnaires in a randomized trial of smoking cessation. Nicotine Tob Res. 2006 Dec;8 Suppl 1(Suppl 1):S49-57. doi: 10.1080/14622200601045367. PMID 17491171
- [Result] Graham AL, Papandonatos GD. Reliability of internet- versus telephone-administered questionnaires in a diverse sample of smokers. J Med Internet Res. 2008 Mar 26;10(1):e8. doi: 10.2196/jmir.987. PMID 18364345
- [Result] Graham AL, Cobb NK, Papandonatos GD, Moreno JL, Kang H, Tinkelman DG, Bock BC, Niaura RS, Abrams DB. A randomized trial of Internet and telephone treatment for smoking cessation. Arch Intern Med. 2011 Jan 10;171(1):46-53. doi: 10.1001/archinternmed.2010.451. PMID 21220660
- [Result] Graham AL, Papandonatos GD, Kang H, Moreno JL, Abrams DB. Development and validation of the online social support for smokers scale. J Med Internet Res. 2011 Sep 28;13(3):e69. doi: 10.2196/jmir.1801. PMID 21955465
- [Result] Graham AL, Chang Y, Fang Y, Cobb NK, Tinkelman DS, Niaura RS, Abrams DB, Mandelblatt JS. Cost-effectiveness of internet and telephone treatment for smoking cessation: an economic evaluation of The iQUITT Study. Tob Control. 2013 Nov;22(6):e11. doi: 10.1136/tobaccocontrol-2012-050465. Epub 2012 Sep 25. PMID 23010696
- [Result] Cobb CO, Niaura RS, Donaldson EA, Graham AL. Quit now? Quit soon? Quit when you're ready? Insights about target quit dates for smoking cessation from an online quit date tool. J Med Internet Res. 2014 Feb 17;16(2):e55. doi: 10.2196/jmir.3086. PMID 24534139
- [Result] Cobb CO, Graham AL. Use of non-assigned interventions in a randomized trial of internet and telephone treatment for smoking cessation. Nicotine Tob Res. 2014 Oct;16(10):1289-97. doi: 10.1093/ntr/ntu066. Epub 2014 May 8. PMID 24812022
- [Result] Graham AL, Papandonatos GD, Cobb CO, Cobb NK, Niaura RS, Abrams DB, Tinkelman DG. Internet and Telephone Treatment for smoking cessation: mediators and moderators of short-term abstinence. Nicotine Tob Res. 2015 Mar;17(3):299-308. doi: 10.1093/ntr/ntu144. Epub 2014 Aug 25. PMID 25156528
- [Result] Graham AL, Papandonatos GD, Erar B, Stanton CA. Use of an online smoking cessation community promotes abstinence: Results of propensity score weighting. Health Psychol. 2015 Dec;34S(0):1286-95. doi: 10.1037/hea0000278. PMID 26651470
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569